CLINICAL TRIAL: NCT03375515
Title: Patient Controlled Analgesia (PCA) vs Non-PCA Intravenous Hydromorphone Titration for Severe Cancer Pain: A Prospective, Randomized, Controlled, Multi-center, Phase III Trial
Brief Title: PCA vs Non-PCA Intravenous Hydromorphone Titration for Severe Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMORCT09-1
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2020-04

CONDITIONS: Cancer Pain
Keywords: hydromorphone titration
MeSH Terms: conditions — Cancer Pain | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCA IV Hydromorphone titration (Experimental): PCA titration using programmable pump: bolus hydromorphone at 0.5mg (for opioid intolerance) or hydromorphone dose equivalent to 10% to 20% of the total opioid taken in the previous 24 hours with a lockout time 15 min (for opioid tolerance) was administered by the patients educated. No basal infusion was set in the pump.Repeated assessment of NRS score with a interval of 15 minutes until stable pain control. Then Repeated assessment of NRS score with a interval of 1 hour. The titration will be done on the patient's request (manipulation by the patient himelf/herself) in 24hrs.
  Interventions: Drug: Hydromorphone; Device: PCA pump
- non-PCA IV Hydromorphone titration (Active Comparator): Non-PCA titration administered by a nurse or clinician: Initial hydromorphone doses were same with PCA titration. Repeated assessment of NRS score with a interval of 15 minutes until stable pain control. Then Repeated assessment of NRS score with a interval of 1 hour. The dose of hydromorphone increased by 50%-100% if pain unchanged or increased, or repeat same dose if pain decrease to 4-6. The titration will be done on the patient's request (manipulation by a nurse) in 24hrs.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — 1. For opioid-intolerant patients: continuous infusion of hydromorphone 0 mg per hour, and a demand dose of 0.5 mg with a lockout interval of 15 minutes.
  2. For opioid-tolerant patients: basal rate 0 mg per hour, and a demand dose of 10% of the hydromorphone dose equivalent to the total opioid taken in the previous 24 hrs with a lockout interval of 15 minutes.
Device: PCA pump — 1. For opioid-intolerant patients: initial dose 0.5 mg intravenous hydromorphone.
  2. For opioid-tolerant patients: intravenous hydromorphone with a initial dose equivalent to 10%(5-15%) of the total opioid taken in the previous 24 hrs.
  Arms: PCA IV Hydromorphone titration

SUMMARY:
A large number of studies have shown that patients feel more satisfied with hydromorphone in the pain management. and a systematic review found that hydromorphone may be better suited than morphine for titration of acute analgesia. However, current researches on intravenous opioid titration for cancer pain such as hydromorphone are relatively insufficient in China. Therefore, a prospective, multi-center, randomized controlled study is conducted to assess the efficacy and safety of comparing patient-controlled analgesia (PCA) versus non-PCA intravenous hydromorphone titration for severe cancer pain.

DETAILED DESCRIPTION:
The opioid dose for individual with cancer pain to provide adequate relief of pain with an acceptable degree of side effects is variable. Opioid titration is a process to obtain the tailored dose. Conventional titration is administered by a clinician or nurse. PCA is that patients control cancer pain by self-administration of intravenous opioids using programmable pump. The aim of our study is to evaluate the efficacy of PCA titration versus conventional titration intravenously for severe cancer pain (10-point numerical rating scale, NRS ≥ 7). Injectable Hydromorphone was selected as pharmaceutical analgesics, which works as well as morphine and oxycodone and had similar side effects.

ELIGIBILITY:
Inclusion Criteria:

1. With written informed consent signed voluntarily by patients themselves.
2. Cancer patients aged 18-70 years old.
3. Patients with cancer pain more than or equal to NRS 7 during previous 24 hours.
4. Patients who will not be treated with radiotherapy within 7 days prior to randomization and during study.
5. Patients who need chemotherapy, long term administration of hormone, targeted therapy, or bisphosphonates therapy should undergo a stable anti- tumor therapy prior to randomization.
6. Patients or his/her caregivers who are able to fill out the questionnaire forms.
7. Ability to correctly understand and cooperate with medication guidance of doctors and nurses.
8. Without a history of anaphylaxis of narcotic drugs.
9. Without psychiatric problems.
10. ECOG performance status ≤3.
11. Not participated in another drug clinical trial within one month before inclusion（including hydromorphone）.

Exclusion Criteria:

1. Patients diagnosed with non-cancer pain or unexplained pain.
2. Patients suffered with post-op pain.
3. Patients having paralytic ileus.
4. Patients who have hypersensitivity to hydromorphone.
5. There are abnormal lab results, with obvious clinical significance, such as the creatinine ≥ 2 fold of upper limit of normal value, or ALT or AST ≥ 2.5 fold of upper limit of normal value (≥ 5 fold,to the patients with liver metastasis or primary liver cancer), or liver function of Child C grade.
6. Patients having a incoercible Nausea and vomiting.
7. Monoamine oxidase inhibitor (MAOI) was administrated two week before randomization.
8. Patients who are pregnant or lactating,who plans to be pregnant within one month after the trial（including male）.
9. Patients who are opioid abuse.
10. Patients who are alcohol abuse.
11. Patients who are cognitive dysfunction.
12. Patients having a severe psychotic depression.
13. Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unable to participate in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
The time of successful titration in 24 hours | In 24 hours
  The satisfied pain control was defined NRS pain score ≤ 3 at rest in at least 2 consecutive assessment (15 minutes interval). The time needed to successful titration was extended to achieve satisfied pain control again if NRS pain score ≥ 7 after satisfied pain control within 24 hours. The failure of successful titration was defined that satisfied pain control does not achieve within 24 hours.

SECONDARY OUTCOMES:
The percentage of patients titrated successfully within 60 minutes | Up to 60 minutes
  The percentage of patients who titrated successfully within 60 minutes
The percentage of patients titrated successfully within 24 hours | Up to 24 hours
  The percentage of patients who titrated successfully within 24 hours
The mean NRS pain score of 24 hours | Up to 24 hours
  The Numerical Rating Scale (NRS) is used to assess the severity of pain. The scale represents pain levels in 0-10 numbers, with 0 indicating no pain and 10 indicating the most severe pain. Ask the patient to choose the number that best represents his or her pain level, or ask the patient to ask: How severe is participant's pain? The health care provider selects the appropriate number based on the patient's description of the pain. 1-3 points indicate mild pain, 4-6 points indicate moderate pain, and 7-10 points indicate severe pain. "The mean NRS pain score of 24 hrs" is defined as the sum of the scores within 24 hours divided by the number of evaluations within 24 hours.
The total dose of hydromorphone titrated from start of titration to TST | Up to 24 hours
  The total dose of hydromorphone titrated from start of titration to TST
The total dose of hydromorphone titrated within 24 hrs | Up to 24 hours
  The total dose of hydromorphone titrated within 24 hrs
Improvement of patient symptoms | Up to 24 hours
  The change from baseline in questionnaire: Chinese version of the Edmonton Symptom Assessment System
Adverse Events | Up to 7 days
  treatment-related Adverse Events:

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, Study Director — Fujian Cancer Hospital
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No